CLINICAL TRIAL: NCT03461705
Title: Derivation and Validation of a Novel Adenosine-independent Index of Coronary Artery Stenosis Severity Resting Flow Reserve
Brief Title: Novel Adenosine-independent Index of Coronary Artery Stenosis Severity Resting Flow Reserve
Acronym: RFR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After 5 patients, realized that the standard deviation of the measurements in real life was higher than the calculated difference.
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Ajay Kirtane, Associate Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAR4732
Record Dates: First submitted 2018-02-22; First posted 2018-03-12 (Actual); Results first posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Coronary; Ischemic
Keywords: Coronary Artery Stenosis; Stenosis; Resting Flow Reserve (RFR); Volcano Verrata Pressure Wire
MeSH Terms: conditions — Ischemia; Coronary Stenosis; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Primary (Experimental): All patients who are referred for coronary angiography and require physiological assessment of intermediate lesions will have both RFR and iFR measured during their standard of care procedure. Both the RFR wire (St. Jude Medical (SJM) Aeris Pressure Wire System) and iFR (Volcano Verrata Pressure Wire) wire will be advanced across the lesion with the sensor located at least 3 cm distal from the lesion.
  Interventions: Device: Volcano Verrata Pressure Wire; Device: St. Jude Medical (SJM) Aeris Pressure Wire System

INTERVENTIONS:
Device: Volcano Verrata Pressure Wire — Steerable guidewire with a pressure transducer mounted 3cm proximal to the tip. The guidewire has a diameter of 0.014".
  and is packaged preconnected to the connector with a torque device to facilitate navigation through the vasculature.
  Other Names: iFR Wire
Device: St. Jude Medical (SJM) Aeris Pressure Wire System — The pressure wire is a 0.014'' guidewire with a pressure and temperature sensor integrated into the tip to enable measurements of physiological parameters.
  Other Names: RFR Wire

SUMMARY:
This study will enroll patients who are referred for coronary angiography and require physiological assessment to see if the lesion can be treated as per the local standard of care. Approximately 92 participants will be enrolled. There are no follow up visits required so participation in this study will end when subjects are discharged from the hospital.The study will be comparing the resting flow reserve against the instantaneous wave-free ratio (iFR) and fractional flow reserve. All these tests offer a way to image a legion and determine if it is suitable to be treated. FFR measures the pressure differences across (narrowed coronary arteries usually due to atherosclerosis), iFR's are performed during cardiac catheterisation (angiography) using invasive coronary pressure wires which are placed in the arteries of the heart that are to be assessed and the Resting flow reserve looks at the maximum increase in blood flow through the coronary arteries above the normal resting volume.

DETAILED DESCRIPTION:
Fractional flow reserve (FFR) measurement by under hyperemic conditions has become the invasive gold standard for determining the physiologic extent of cardiac ischemia, and which has been validated in several clinical outcomes studies as a way of optimizing case selection for percutaneous coronary intervention (PCI). More recently in two large-scale randomized controlled trials using a non-hyperemic resting measurement, the instantaneous wave free ratio (iFR) showed non-inferiority in major adverse cardiovascular events (MACE) comparing iFR to FFR for physiological assessment of moderate coronary stenosis. FFR is calculated as the ratio of the distal coronary pressure to the aortic pressure (Pd/Pa) during maximal micro-circulatory relaxation. iFR is a diagnostic tool used to assess whether a stenosis is causing a limitation of blood flow in coronary arteries with subsequent ischemia. iFR is performed during cardiac catheterization (angiography) using invasive coronary pressure wires which are placed in the coronary arteries that are to be assessed. The iFR negates the time averaging and administration of vasodilators necessary for FFR by identifying from the resting pressure waveform a period when the native microcirculatory resistance is constant and minimized in diastole. The study is looking at the accuracy and precision of a novel adenosine-independent index of coronary artery stenosis, the resting flow reserve, against the instantaneous wave-free ratio and fractional flow reserve.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patient provides signed written informed consent before any study-specific procedure.
3. Undergoing coronary angiography, for silent ischemia, stable angina, acute coronary syndrome, or other acceptable indication per the local standard of care.
4. Angiographically 40%-90% stenosis present in at least one native coronary artery.
5. Undergoing physiological assessment for standard clinical or diagnostic indications

Exclusion Criteria:

1. Aorto-ostial lesion location within 3 mm of the aorta junction (both right and left).
2. Left main stenosis
3. Vessel(s) and lesion(s) not amenable for percutaneous coronary intervention (PCI) , for example diffuse disease.
4. Saphenous vein graft, chronic total occlusion
5. Haemodynamic instability at the time of intervention (heart rate<50 beats per minute, systolic blood pressure <90mmHg), balloon pump
6. Currently participating in another clinical study that interferes with study results.
7. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure.
8. Any other medical condition that in the opinion of the investigator will interfere with patient safety or study results.
9. High degree A-V block, sinus node disease.
10. Asthma/Chronic obstructive pulmonary disease (COPD) with active wheeze
11. Known hypersensitivity to adenosine
12. ST-Elevation Myocardial Infarction (STEMI) within 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Kirtane, MD, Principal Investigator — CUMC
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary: All patients who are referred for coronary angiography and require physiological assessment of intermediate lesions will have both RFR and iFR measured during their standard of care procedure. Both the RFR wire (St. Jude Medical (SJM) Aeris Pressure Wire System) and iFR (Volcano Verrata Pressure Wire) wire will be advanced across the lesion with the sensor located at least 3 cm distal from the lesion.
  Volcano Verrata Pressure Wire: Steerable guidewire with a pressure transducer mounted 3cm proximal to the tip. The guidewire has a diameter of 0.014".
  and is packaged preconnected to the connector with a torque device to facilitate navigation through the vasculature.
  St. Jude Medical (SJM) Aeris Pressure Wire System: The pressure wire is a 0.014'' guidewire with a pressure and temperature sensor integrated into the tip to enable measurements of physiological parameters.
Period: Overall Study
Arm/Group | Primary
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Primary
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 5
Referred for Coronary Angiography [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage Agreement Between Mean RFR and iFR Measurements
Description: Mean RFR measurements will be compared against mean iFR measurements to determine if there is an agreement between RFR and iFR for detection of ischemia.
Time Frame: During procedure
Population: After 5 patients, investigators realized that the standard deviation of the measurements in real life was higher than the calculated difference that could have existed between the two different measurement techniques and therefore did not collect or analyze the data for the 5 subjects (out of a target of 92).
Arm/Group | Primary
Number analyzed (Participants) | 0

2. Secondary Outcome: Lesion Classification (FFR≤/>0.80) by RFR
Time Frame: During procedure
Population: as for outcome 1
Arm/Group | Primary
Number analyzed (Participants) | 0

3. Secondary Outcome: Lesion Classification (FFR≤/>0.80) by iFR
Time Frame: During procedure
Population: as for outcome 1
Arm/Group | Primary
Number analyzed (Participants) | 0

4. Secondary Outcome: Pressure Drift of RFR
Time Frame: During procedure
Population: as for outcome 1
Arm/Group | Primary
Number analyzed (Participants) | 0

5. Secondary Outcome: Pressure Drift of iFR
Time Frame: During procedure
Population: Since only 5 out of 92 were treated, data was not systematically collected and analysis was not performed.
Arm/Group | Primary
Number analyzed (Participants) | 0

6. Secondary Outcome: Measurement Reproducibility for RFR
Description: Reproducibility of RFR will be tested against iFR. Reproducibility will be measured by comparing the measure of RFR (minimal ratio of distal coronary pressure/aortic pressure) at time point 1 versus time point 2 against iFR (minimal ratio of distal coronary pressure/aortic pressure during the wave-free period of diastole) at time point 1 versus time point 2.
Time Frame: During procedure
Population: as for outcome 1
Arm/Group | Primary
Number analyzed (Participants) | 0

7. Secondary Outcome: Measurement Reproducibility for iFR
Description: Reproducibility of iFR will be tested against RFR. Reproducibility will be measured by comparing the measure of iFR (minimal ratio of distal coronary pressure/aortic pressure during the wave-free period of diastole) at time point 1 versus time point 2 against RFR (minimal ratio of distal coronary pressure/aortic pressure) at time point 1 versus time point 2.
Time Frame: During procedure
Population: as for outcome 1
Arm/Group | Primary
Number analyzed (Participants) | 0

8. Secondary Outcome: Ability to Advance to the Target Lesion and Measure RFR and iFR
Description: Percentage of technical failure due to the inability to deliver the wire and measure out of total number of all procedures
Time Frame: During procedure
Population: as for outcome 1
Arm/Group | Primary
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day of the procedure.
Arm/Group | Primary
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
The standard deviation of the measurements in real life was higher than the calculated difference that could have existed between the two different measurement techniques so study halted early and data was not collected and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT03461705/Prot_SAP_000.pdf